CLINICAL TRIAL: NCT04453800
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Sofadil for Injection in the Treatment of Acute Ischemic Stroke
Brief Title: The Efficacy and Safety of Sofadil for Injection in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUTH2017013
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Sofadil; Acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Contraceptives, Oral

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study will be conducted in a double-blind form. The clinical research team participating in the study will be divided into two groups: blind and non-blind members, strictly ensuring that researchers and subjects are blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A ：low dose sofadil (Experimental): 500mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 250mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Interventions: Drug: sofadil【Neu2000KW】
- Group B: Medium dose group (Experimental): 750mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 500mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Interventions: Drug: Sofadil
- Group C: high dose group (Experimental): 1500mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 500mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Interventions: Drug: Sofadil
- Group D: placebo group (Placebo Comparator): Saline was administered intravenously
  Interventions: Other: placebo

INTERVENTIONS:
Drug: sofadil【Neu2000KW】 — 500mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 250mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Other Names: low dose
  Arms: Group A ：low dose sofadil
Drug: Sofadil — 750mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 500mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Other Names: Medium dose
  Arms: Group B: Medium dose group
Drug: Sofadil — 1500mg Intravenous infusion of sofadil starting at 500mg was 500ml，followed by nine intravenous infusions, each 500mg infusion with 250ml sofadil for 5 days, and each interval is 12 hours
  Other Names: high dose
  Arms: Group C: high dose group
Other: placebo — Saline was administered intravenously
  Arms: Group D: placebo group

SUMMARY:
To evaluate the efficacy and safety of sofadil injection in the treatment of acute ischemic stroke

DETAILED DESCRIPTION:
The limited therapeutic time window for neuroprotection has prevented all clinical trials using NMDA receptor antagonists in subjects with ischemic stroke from showing efficacy. In animal models of ischemic stroke, antioxidants showed a longer neuroprotective time window than NMDA receptor antagonists, and also showed therapeutic potential in clinical trials in subjects with ischemic stroke. Sophadil showed good neuroprotective effects against NMDA and free-radical mediated cell death, NR2B-selectivity, moderate NMDA receptor antagonism, and effective cellular osmotic antioxidant activity even at nanoscale molarity. Non-clinical and phase I human clinical studies have shown that Sofadil is helpful in treating ischemic stroke subjects with better efficacy and therapeutic time windows. So we designed the clinical trial to evaluate the efficacy and safety of sofadil injection in the treatment of acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

* The target population is 35-75 years old, regardless of gender;
* within 6h of onset, ischemic stroke of the internal carotid artery system;
* Neurological deficits, including limb weakness, with acute brain injury (NIHSS score) (4-22 points), or NIHSS item 5 upper limb or 6 lower limb score ≥2 points;
* Be able to initiate study treatment within 6 hours of onset of symptoms or within 6 hours of last appearing normal (6 hours after sleep in subjects with ischemic stroke who developed during sleep) and complete post-onset CT examination prior to study treatment;
* Obtain the informed consent signed by the subject or the subject's legal representative;
* MRS score before onset was 0~1;
* Patients with no history of myocardial infarction within 3 months;
* Centerless, liver, kidney and lung dysfunction;
* No hemorrhagic disease within 3 months;
* No blood system diseases.

Exclusion Criteria:

* Any contraindications to CT or MRI (such as metal implants such as pacemaker, claustrophobia, etc
* Stroke caused by posterior circulation ischemia, or TIA;
* Acute intracranial hemorrhage, intracranial tumor, subarachnoid hemorrhage, encephalitis or other non-acute ischemic stroke (onset less than 6 hours), intracranial arteriovenous malformations;
* Patients who plan to undergo endovascular treatment, such as mechanical thrombectomy, stenting or arteriovenous bridging, within 6 hours after onset;
* Pregnant or lactating women. Note: The blood pregnancy test for fertile women before randomization must be negative and appropriate contraception should be used at least 3 weeks before randomization until 7 days after study drug infusion
* A pre-existing medical, neurological or psychiatric disorder that confuses neurological, functional or imaging assessments, such as persistent injury from previous ischemic stroke;
* Patients with malignant tumors or other critical diseases;
* Having a history of epilepsy or having epileptiform symptoms at the onset of stroke;
* Previous history of intracranial hemorrhage;
* Patients with previous hypotension or blood pressure of less than 90/60mmhg measured for 3 consecutive times;
* Patients with severe injuries and surgical history within 3 months;
* People with consciousness disorder can be defined as "NIHSS score Ia ≥2 points";
* Bradycardia with complete atrioventricular block;
* According to the New York heart association (NYHA) grade of cardiac function, cardiac function rating above Ⅱ level, a history of congestive heart failure (CHF).
* Patients with primary liver and kidney diseases, AST or ALT twice as high as the normal upper limit, serum creatinine >2.0 mg/dL or >176.8 mol/L;
* Where the INR is greater than 1.7 or where an oral anticoagulant is currently used, except aspirin, clopidogrel, subcutaneous heparin or Wartamine;
* Patients with bleeding tendency diseases (such as hemophilia), and partial thromboplastin time (PTT) is more than 3 times of the normal upper limit;
* Having a current drug or alcohol problem or experience;
* Has the experience of allergic reaction to the research drugs or drugs with similar chemical structure;
* Participated in other clinical trials or clinical study participants within 3 months before the start of this study;
* The researcher considered it inappropriate to participate in the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a NIHSS score | 14±2 days of treatment
  Proportion of subjects with a NIHSS score of 0 ~ 1 or 4 or more points less than baseline NIHSS at 14±2 days of treatment

SECONDARY OUTCOMES:
Changes in NIHSS score | at 14±2, 30±2, and 90±7 days after treatment compared to baseline
  Changes in NIHSS score at 14±2, 30±2, and 90±7 days after treatment compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, MD.PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Dongsheng Fan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No